CLINICAL TRIAL: NCT04812262
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Dose Study to Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DD01 in Overweight/Obese Subjects With T2DM and NAFLD
Brief Title: A Phase 1 Study of DD01 in Overweight/Obese Subjects With T2DM and NAFLD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuraly, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DD01-DN-1
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Overweight and Obesity; Type2 Diabetes; NAFLD
Keywords: Liver Disease
MeSH Terms: conditions — Overweight; Obesity; Non-alcoholic Fatty Liver Disease; Liver Diseases

STUDY DESIGN:
Intervention Model Description: Part A - Cohorts A1, A2, A3, A4, A5, A6, A7 & A8 Part B - Cohorts B2, B3, B4, B5, B6, B7 & B8
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Group A1 - Single Ascending Dose (Experimental): DD01 Dose 1 (N=6) Placebo (N=2) Subcutaneous injection
  Interventions: Drug: DD01; Drug: Placebo
- Group A2, Single Ascending Dose (Experimental): DD01 Dose 2 (N=6) Placebo (N=2) Subcutaneous injection
  Interventions: Drug: DD01; Drug: Placebo
- Group A3, Single Ascending Dose (Experimental): DD01 Dose 3 (N=6) Placebo (N=2) Subcutaneous injection
  Interventions: Drug: DD01; Drug: Placebo
- Group A4, Single Ascending Dose (Experimental): DD01 Dose 4 (N=6) Placebo (N=2) Subcutaneous injection
  Interventions: Drug: DD01; Drug: Placebo
- Group B2 - Multiple Ascending Dose (Experimental): DD01 Dose 2 (N=6) Placebo (N=2) Subcutaneous injection once weekly for 4 weeks
  Interventions: Drug: DD01; Drug: Placebo
- Group B3 - Multiple Ascending Dose (Experimental): DD01 Dose 3 (N=6) Placebo (N=2) Subcutaneous injection once weekly for 4 weeks
  Interventions: Drug: DD01; Drug: Placebo
- Group B4 - Multiple Ascending Dose (Experimental): DD01 Dose 4 (N=6) Placebo (N=2) Subcutaneous injection once weekly for 4 weeks
  Interventions: Drug: DD01; Drug: Placebo
- Group B5 - Multiple Ascending Dose (Experimental): DD01 Dose 4 (N=6) Placebo (N=2) Subcutaneous injection once weekly for 4 weeks
  Interventions: Drug: DD01; Drug: Placebo
- Group B6 - Multiple Ascending Dose (Experimental): DD01 Dose 4 (N=6) Placebo (N=2) Subcutaneous injection once weekly for 4 weeks
  Interventions: Drug: DD01; Drug: Placebo
- Group A5, Single Ascending Dose (Experimental): DD01 Dose 4 (N=6) Placebo (N=2) Subcutaneous injection
  Interventions: Drug: DD01; Drug: Placebo
- Group A6, Single Ascending Dose (Experimental): DD01 Dose 4 (N=6) Placebo (N=2) Subcutaneous injection
  Interventions: Drug: DD01; Drug: Placebo
- Group A7, Single Ascending Dose (Experimental): DD01 Dose 4 (N=6) Placebo (N=2) Subcutaneous injection
  Interventions: Drug: DD01; Drug: Placebo
- Group A8, Single Ascending Dose (Experimental): DD01 Dose 4 (N=6) Placebo (N=2) Subcutaneous injection
  Interventions: Drug: DD01; Drug: Placebo
- Group B7 - Multiple Ascending Dose (Experimental): DD01 Dose 4 (N=6) Placebo (N=2) Subcutaneous injection once weekly for 4 weeks
  Interventions: Drug: DD01; Drug: Placebo
- Group B8 - Multiple Ascending Dose (Experimental): DD01 Dose 4 (N=6) Placebo (N=2) Subcutaneous injection once weekly for 4 weeks
  Interventions: Drug: DD01; Drug: Placebo

INTERVENTIONS:
Drug: DD01 — The active of DD01 is a synthetic peptide, administered in a 1mL volume for injection.
Drug: Placebo — Placebo drug of DD01, administered in a 1mL volume for injection

SUMMARY:
This is a Phase 1, first in human (FiH), randomized, double-blind, placebo-controlled, single ascending dose (SAD) and multiple ascending dose (MAD) study to investigate the safety, tolerability, PK and PD of DD01 administered by subcutaneous (SC) injection in overweight/obese subjects with type 2 diabetes (T2DM) and nonalcoholic fatty liver disease (NAFLD).

The study will be conducted in 2 Parts (Part A and B), with up to 8 cohorts included in each part (Part A; Cohorts A1 to A8 and Part B; Cohorts B2 to B8).

DETAILED DESCRIPTION:
Part A (SAD):

In Part A, subjects will receive a single dose of study drug, and the safety and efficacy of DD01 will be evaluated in overweight/obese subjects with T2DM.

Part B (MAD):

In Part B, subjects will receive once-weekly doses of the study drug for 4 weeks, and the safety and efficacy of DD01 will be evaluated in overweight/obese subjects with T2DM and NAFLD.

ELIGIBILITY:
Part A Inclusion Criteria:

* Type 2 diabetes ≥ 12 months.
* Treatment with diet and exercise or metformin monotherapy on stable dose for 3 months prior to screening
* HbA1c ≤ 10%).
* Body Mass Index (BMI) ≥ 25 and ≤ 40.0 kg/m2

Part B Inclusion Criteria

* Type 2 diabetes ≥ 12 months.
* Treatment with diet and exercise or metformin monotherapy on stable dose for 3 months prior to screening
* HbA1c ≤ 10%
* BMI ≥ 30 kg/m2 and ≤ 40.0 kg/m2
* Waist circumference ≤ 57 inches
* Controlled attenuation parameter by FibroScan
* Liver fat fraction ≥ 10% by magnetic resonance imaging (MRI)

Part A Exclusion Criteria:

* History of type 1 diabetes mellitus (T1DM)
* History of acute proliferative retinopathy or maculopathy, severe gastroparesis, and/or severe neuropathy, in particular autonomic neuropathy, as judged by the Investigator.
* Uncontrolled hypertension
* Treatment with antihypertensive medication and statins not stable during the past 2 months prior to screening
* Treatment with thyroid hormones not stable during the past 3 months prior to screening
* History of any weight control treatment, including over-the-counter and herbal medication and supplements, or any medication with a labeled indication for weight loss or weight gain within 3 months prior to screening
* History of surgical treatment for obesity
* History of heart disease
* History of renal disease
* History or current diagnosis of acute or chronic pancreatitis or factors for pancreatitis, such as a history of cholelithiasis (without cholecystectomy) or alcohol abuse
* A history of or active chronic liver disease due to alcohol, auto-immune, HIV, HBV or active HCV-infection or NASH
* History of major depression, anxiety, suicidal behavior or attempts, or other psychiatric disorder requiring medical treatment
* Personal or family history of medullary thyroid carcinoma (MTC) or a genetic condition that predispose to MTC (i.e., multiple endocrine neoplasia type 2)
* Administration of Vaccines/Immunizations within 14 days prior to first dosing or if scheduled during the study. Vaccination for COVID-19 is allowed during the study if a washout period of 5 days after vaccine administration is followed before dosing.
* History of any major surgery within 6 months prior to screening
* Participation in any other clinical interventional study receiving active treatment within 30 days or 5 half-lives prior to screening, whichever is longer
* History of alcohol or illicit drug abuse including marijuana
* Existence of any surgical or medical condition that, in the judgment of the Investigator, might interfere with the investigational product

PART B Exclusion Criteria

* History of type 1 diabetes mellitus (T1DM)
* History of acute proliferative retinopathy or maculopathy, severe gastroparesis, and/or severe neuropathy, in particular autonomic neuropathy, as judged by the Investigator
* Uncontrolled hypertension (treatment with medications must be stable)
* History of any weight control treatment
* History of surgical treatment for obesity
* History of heart disease
* History of renal disease
* Subjects with a history or clinically significant active disease of the gastrointestinal, cardiovascular, hepatic, neurological, renal, pancreatic, immunological, dermatological, endocrine, genitourinary or hematological system.
* History or current diagnosis of acute or chronic pancreatitis
* History of major depression, anxiety, suicidal behavior or attempts, or other psychiatric disorder requiring medical treatment
* History of alcohol or illicit drug abuse including marijuana
* Existence of any surgical or medical condition that, in the judgment of the Investigator, might interfere with the investigational product
* Any history of clinically significant chronic liver disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events and serious adverse events | Part A - 43 days
Number of participants with treatment-related adverse events and serious adverse events (TEAEs) | Part B - 57 days
Number of participants with clinically significant abnormalities in clinical laboratory values | Part A - 43 days
Number of participants with clinically significant abnormalities in clinical laboratory values | Part B - 57 days
Number of participants with clinically significant abnormalities in physical examinations | Part A - 43 days
Number of participants with clinically significant abnormalities in physical examinations | Part B - 57 days
Number of participants with clinically significant abnormalities in vital signs | Part A - 43 days
Number of participants with clinically significant abnormalities in vital signs | Part B - 57 days
Blood Pressure assessed by 24-hour ambulatory blood pressure monitoring (ABPM) | Part A - 43 days
Blood Pressure assessed by 24-hour ambulatory blood pressure monitoring (ABPM) | Part B - 57 days
Heart Rate assessed by 24-hour ambulatory electrocardiography monitoring reader) | Part A - 43 days
Heart Rate assessed by 24-hour ambulatory electrocardiography monitoring reader) | Part B - 57 days
Number of participants with clinically significant abnormalities in 12-lead ECGs | Part A - 43 days
Number of participants with clinically significant abnormalities in 12-lead ECGs | Part B - 57 days

SECONDARY OUTCOMES:
Maximum observed blood/plasma concentration of DD01 | Part A - 43 days
  Maximum observed blood/plasma concentration (Cmax)
Maximum observed blood/plasma concentration of DD01 | Part B - 57 days
  Maximum observed blood/plasma concentration (Cmax)
Time of the maximum observed blood/plasma concentration of DD01 | Part A - 43 days
  Time of the maximum observed blood/plasma concentration (Tmax)
Time of the maximum observed blood/plasma concentration of DD01 | Part B - 57 days
  Time of the maximum observed blood/plasma concentration (Tmax)
Apparent blood/plasma terminal elimination half life of DD01 | Part A - 43 days
  Apparent blood/plasma terminal elimination half life (t1/2)
Apparent blood/plasma terminal elimination half life of DD01 | Part B - 57 days
  Apparent blood/plasma terminal elimination half life (t1/2)
Termination elimination rate constant of DD01 | Part A - 43 days
  Termination elimination rate constant (kel)
Termination elimination rate constant of DD01 | Part B - 57 days
  Termination elimination rate constant (kel)
Apparent total blood/plasma clearance of DD01 | Part A - 43 days
  Apparent total blood/plasma clearance (CL/F)
Apparent total blood/plasma clearance of DD01 | Part B - 57 days
  Apparent total blood/plasma clearance (CL/F)
Apparent volume of distribution of DD01 | Part A - 43 days
  Apparent volume of distribution(Vz/F)
Apparent volume of distribution of DD01 | Part B - 57 days
  Apparent volume of distribution(Vz/F)
Area under the blood/plasma concentration time curve from time zero to the time of the last quantifiable concentration of DD01 | Part A - 43 days
  Area under the blood/plasma concentration time curve from time zero to the time of the last quantifiable concentration (AUC0-t)
Area under the blood/plasma concentration time curve from time zero to the time of the last quantifiable concentration of DD01 | Part B - 57 days
  Area under the blood/plasma concentration time curve from time zero to the time of the last quantifiable concentration (AUC0-t)
Area under the blood/plasma concentration time curve from time zero to 144 hours postdose of DD01 | Part A - 43 days
  Area under the blood/plasma concentration time curve from time zero to 144 hours postdose (AUC0-144)
Area under the blood/plasma concentration time curve from time zero to 144 hours postdose of DD01 | Part B - 57 days
  Area under the blood/plasma concentration time curve from time zero to 144 hours postdose (AUC0-144)
Area under the blood/plasma concentration time curve from time zero to 216 hours postdose of DD01 | Part A - 43 days
  Area under the blood/plasma concentration time curve from time zero to 216 hours postdose (AUC0-216)
Area under the blood/plasma concentration time curve from time zero to 216 hours postdose of DD01 | Part B - 57 days
  Area under the blood/plasma concentration time curve from time zero to 216 hours postdose (AUC0-216)
Area under the blood/plasma concentration time curve from time zero to 168 hours postdose of DD01 | Part B - 57 days
  Part B only: Area under the blood/plasma concentration time curve from time zero to 168 hours postdose (AUC0-168)
Number of participants with antidrug antibodies (ADAs) | Part A - 43 days
Number of participants with antidrug antibodies (ADAs) | Part B - 57 days

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Prosciento, Chula Vista, California
  - Southwest General Healthcare Center, Fort Myers, Florida
  - Combined Research Orlando, Orlando, Florida
- FDI Clinical Research, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No